CLINICAL TRIAL: NCT03271879
Title: The Effect of Empagliflozin Versus Placebo on the Rate of Arrhythmic Events in Heart Failure Patients
Brief Title: Empagliflozin Versus Placebo on the Rate of Arrhythmic Events in Heart Failure Patients
Acronym: ERA-HF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 605-16
Record Dates: First submitted 2017-07-30; First posted 2017-09-05 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure; Diabetes Mellitus; Arrythmia
Keywords: Diabetes; Heart; Arrhythmia
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Patients will receive study drug: empagliflozin or placebo for an exposure period of up to 16 weeks - at the two treatment periods in a crossover design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin at a dose of 10 mg/day (Active Comparator): Patients will be treated with 10mg Empagliflozin once daily for 8 weeks. Patient glucose levels will be monitored based on home monitoring during the treatment period.
  Interventions: Drug: Empagliflozin at a dose of 10 mg/day
- Placebo (Placebo Comparator): Patients will be treated with Placebo once daily for 8 weeks. Patient glucose levels will be monitored based on home monitoring during the treatment period.
  Interventions: Drug: Empagliflozin at a dose of 10 mg/day

INTERVENTIONS:
Drug: Empagliflozin at a dose of 10 mg/day — Comparing empagliflozin versus placebo on the ventricular arrhythmia burden. This study encompass 4 periods for each study subject: screening period of 8 weeks, first treatment period of 8 weeks, washout period of 4 weeks and a second treatment period of 8 weeks in a cross-over design
  Other Names: JARDIANCE at a dose of 10mg/day

SUMMARY:
Empagliflozin treatment in high cardiovascular risk patients has been shown to have a relatively rapid powerful capability in reducing cardiovascular mortality. Among the suggested mechanisms mediating this effect of empagliflozin, anti-arrhythmic effect (AAE) has the highest potential to translate into a rapid clinical beneficial effect on cardiovascular mortality, while other mechanisms are known to have a lag in their clinical effect based on data from previous studies. Based on this assumption, the study driving hypothesis is that the effect of empagliflozin on the rate of cardiovascular death may be mediated by a direct effect on the risk for arrhythmic events (via a direct or an indirect effect on the myocardium). The current study aims at assessing the effect of empagliflozin on arrhythmias in diabetic patients with HF with reduced ejection fraction and relatively high arrhythmic burden. The objective of the current study is to demonstrate the effect of empagliflozin compared to placebo on the rate of ventricular arrhythmic events in type 2 diabetes patients with heart failure with reduced ejection fraction and high risk arrhythmic profile.

DETAILED DESCRIPTION:
Background and rationale: Empagliflozin is an orally available inhibitor of the sodium-glucose co-transporter 2 (SGLT-2), that promotes enhanced glucose excretion in the urine, thereby lowering blood glucose concentrations in patients with type 2 diabetes mellitus (T2DM). The EMPA-REG OUTCOME study demonstrated a significant reduction in both heart failure hospitalization and cardiovascular death in type 2 diabetes patients with high risk for cardiovascular events. A potential mechanism underlying the pleiotropic and explaining the remarkable early reduction in cardiovascular mortality may be related to the effect of empagliflozin on arrhythmic events.

Multiple potential mechanisms have been suggested to mediate the positive cardiovascular effect of empagliflozin (altered cardiomyocyte metabolism, anti-arrhythmic effect, improved glycemic control, positive effect on myocardial contractility).

Ventricular arrhythmias and the associated sudden cardiac death (SCD) is the leading cause of mortality in patients with heart failure. The risk for the occurrence of SCD in heart failure patients is closely related to the etiology (ischemic versus non-ischemic) and the left ventricular EF. The introduction of defibrillation therapy for primary prevention of SCD in HF patients has revolutionized the field during the last 2 decades. Nevertheless, ventricular arrhythmias remain a major cause of mortality for HF patients given the limited ability for risk stratification, and the dreadful prognosis associated with ventricular arrhythmias treated by defibrillation therapy. The burden of premature ventricular Complexes (PVCs) has been shown as an independent risk factor for ventricular tachyarrhythmia and SCD for healthy, ischemic and heart failure patients (with and without resynchronization and/or defibrillator therapy). Anti-arrhythmic drugs (AAD) are efficient in suppressing the occurrence of PVCs but for certain drugs, the associated with profile of adverse events and cardiotoxicity may paradoxically increase the rate of sudden cardiac death as learned by the remarkable CAST study. Be that as it may, easily suppressed PVC burden (without the associated adverse profile of AADs) has been suggested to correlate with reduction of the likelihood for SCD. Furthermore, the growing field of PVC ablation has been shown to have beneficial effect on cardiac function and the risk for ventricular arrhythmia. In summary, PVC suppression, a once neglected strategy, is now considered a promising strategy for evaluating the effect of therapeutic strategies on the risk for SCD.

Empagliflozin treatment in high cardiovascular risk patients has been shown to have a relatively rapid powerful capability in reducing cardiovascular mortality. Among the suggested mechanisms mediating this effect of empagliflozin, anti-arrhythmic effect (AAE) has the highest potential to translate into a rapid clinical beneficial effect on cardiovascular mortality, while other mechanisms are known to have a lag in their clinical effect based on data from previous studies. Based on this assumption, the study driving hypothesis is that the effect of empagliflozin on the rate of cardiovascular death may be mediated by a direct effect on the risk for arrhythmic events (via a direct or an indirect effect on the myocardium). The current study aims at assessing the effect of empagliflozin on arrhythmias in diabetic patients with HF with reduced EF and relatively high arrhythmic burden.

Study Objectives The objective of the current study is to demonstrate the effect of empagliflozin compared to placebo on the rate of ventricular arrhythmic events in type 2 diabetes patients with heart failure with reduced ejection fraction and high risk arrhythmic profile.

Primary endpoint:

The primary endpoint is the burden of premature ventricular complexes, defined as the PVCs percentage of all beats in a pre-specified period captured on implantable cardioverter-defibrillator ( ICD ) or CRTD/P device.

Secondary endpoint:

1. The number of non-sustained ventricular tachycardia (NSVT) episodes.
2. A composite cumulative endpoint of ventricular arrhythmia load (number of: sustained ventricular tachycardia, ventricular fibrillation, antitachycardia pacing (ATP) or delivery of shock therapy episodes.
3. The change in blood level of NT-Pro Brain Natriuretic peptide (BNP) from baseline to the end of any of the treatment periods.
4. The change in Left ventricular end diastolic diameter on echocardiography from baseline to the end of any of the treatment periods.
5. The change in left ventricular ejection fraction (EF) on echocardiography from baseline to the end of any of the treatment periods.
6. Safety endpoints (as detailed bellow).

Study Design:

The present study is a randomized, prospective, controlled, double blind, cross-over, pairwise, add on standard therapy, event driven study, comparing empagliflozin versus placebo on the ventricular arrhythmia burden in a blocked randomization stratified by ischemic versus non-ischemic cardiomyopathy and PVC burden at screening of< or > to 4%. Potential study subjects will sign an informed consent prior to undergoing any study related procedure. Number of patients to be enrolled is 128.

This study encompass 4 periods for each study subject: screening period of 8 weeks, first treatment period of 8 weeks, washout period of 4 weeks and a second treatment period of 8 weeks. Expected duration of subject participation is 6-7 months.

Duration of study:

The duration of the treatment period is approximately 6 months. This time span is required for completing the therapy and determining the safety profile of the drug combination and the response rate.

Estimated accrual duration: 12 months. Estimated total trial duration: 18 months (for each center).

ELIGIBILITY:
Inclusion Criteria:

1. Heart failure patients with reduced ejection fraction (EF≤40%) as assessed by echocardiographist least 6 months prior to recruitment and NYHA Class≥2
2. Patients implanted with ICD, CRTD/S or CRTP devices that are capable of recording the PVC burden and implanted ≥ 2 months prior to recruitment.
3. High risk for arrhythmic events at baseline identified by either PVC burden ≥0.5% or ≥2 events of non sustained VT or ≥1 event of sustained ventricular tachycardia or need for anti-tachycardia pacing or defibrillation therapy, during a period of 2 months prior to recruitment.
4. Diagnosis of type 2 diabetes mellitus prior to informed consent
5. HbA1c≥7% and ≤12%.
6. Signed and dated written informed consent by date of Visit 1 in accordance with GCP legislation

   -

Exclusion Criteria:

1. Evidence of ICD malfunction.
2. Past exposure to SGLT2 inhibitors.
3. Uncontrolled diabetes with HbA1c>12% or glucose >240 mg/dL after an overnight fast.
4. Liver abnormalities defined by serum levels of alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase above 3 x upper limit of normal.
5. Planned cardiac procedure within 3 months.
6. Prior MI in the last 40 days.
7. Calculated eGFR< 45ml/min/1.73m2 as determined by the MDRD formula GFR (mL/min/1.73 m2) = 175 × (Scr)-1.154 × (Age)-0.203 × (0.742 if female) × (1.212 if African American)
8. BMI>50
9. Medical History of active cancer in the last 2 years. Exceptions include the following: Basal cell carcinoma of the skin, Squamous cell carcinoma of the skin, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b).
10. History of recurrent UTIs or genital infections
11. Systolic blood pressure< 90 mmHg.
12. Alcohol or drug abuse within 3 months of informed consent.
13. Pre-menopausal women (last menstruation <+ 1 year prior to informed consent) who:

    * - are nursing or pregnant or
    * - are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include tubal ligation, transdermal patch, intra uterine devices/systems, oral, implantable or injectable contraceptives, sexual abstinence, double barrier method and vasectomised partner.
14. Intake of an investigational drug in another trial within 30 days prior to intake of study medication in this trial or participating in another trial involving an investigational drug and/or follow-up

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2018-02-15 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the burden of premature ventricular complexes, defined as the PVCs percentage of all beats in a pre-specified period captured on ICD or CRTD/P device | Time frames include the time frame between visit 2 (on day 56) and visit 3 (on day 112) and that between visit 4 (on day 140) to visit 5 (on day 196)- each period between visits 2 and 3 and visit 4 and 5 contain a time frame of 56 days
  PVCs burden is defined as the PVCs percentage of all beats in a pre-specified period captured on ICD or CRTD/P device. The change in PVC burden between time on treatment arm versus time on placebo will be calculated and serve as the primary endpoint.

SECONDARY OUTCOMES:
Non-sustained ventricular tachycardia (NSVT) | Time frames include the time frame between visit 2 (on day 56) and visit 3 (on day 112) and that between visit 4 (on day 140) to visit 5 (on day 196)- each period between visits 2 and 3 and visit 4 and 5 contain a time frame of 56 days
  This is defined as the number of sustained ventricular tachycardia, and/or ventricular fibrillation, and/or tachycardia pacing (ATP) and/or delivery of shock therapy. All the four parameters will be captured on ICD or CRTD/P device interrogation. Sustained VT and NSVT will be captured as a backup information (in case of ICD or CRTD/P malfunction) on Holter ECG.
NT-Pro-BNP | Time frames include NT-Pro-BNP measurement on the end of visit 3 (on day 112) versus NT-Pro-BNP level at the end of visit 5 (on day 196).
  NT-Pro-BNP Is a plasma level of B-type Natriuretic Peptide used as a blood test for diagnosing and evaluation the presence/severity of heart failure. The change in NT-Pro-BNP will be evaluated as a marker of heart failure severity.
Left ventricular end diastolic diameter | Time frames include left ventricular diastolic diameter measured on the end of visit 3 (on day 112) versus that measured at the end of visit 5 (on day 196).
  End diastolic diameter is defined as the cross-sectional diameter of the left ventricle, including the septum and the posterior thicknesses in diastole.
Left ventricular ejection fraction (EF) | Time frames include EF measured on visit 3 (on day 112) versus that measured at the end of visit 5 (on day 196).
  Ejection fraction is defined as the ratio of the stroke volume to the end-diastolic volume in the left ventricle as performed by echocardiography and expressed by percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Oren Caspi, MD, Principal Investigator — Rambam MC

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared following approval of the submitted research proposal by the researcher applying.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT03271879/Prot_SAP_000.pdf